CLINICAL TRIAL: NCT05388058
Title: Topical Cannabidiol (CBD) for the Treatment of Chemotherapy-Induced Peripheral Neuropathy: A Randomized Placebo-Controlled Pilot Trial
Brief Title: Topical Cannabidiol for the Treatment of Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MC211003; NCI-2022-02479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-011969 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2024-04

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Malignant Solid Neoplasm
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cannabidiol, placebo) (Experimental): Patients apply cannabidiol cream topically to affected areas BID for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.
  Interventions: Drug: Cannabidiol; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo, cannabidiol) (Experimental): Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.
  Interventions: Drug: Cannabidiol; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cannabidiol — Applied topically
  Other Names: CBD; CBD Oil; Epidiolex; GWP42003-P
Drug: Placebo Administration — Applied topically
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares topical cannabidiol to placebo in improving chemotherapy-induced peripheral neuropathy, or painful sensations in your hands or feet due to chemotherapy. Peripheral neuropathy is a nerve problem that causes pain, numbness, tingling, swelling, or muscle weakness in different parts of the body. It usually begins in the hands or feet and gets worse over time. Peripheral neuropathy caused by chemotherapy is called chemotherapy-induced peripheral neuropathy (CIPN). CIPN is commonly seen in patients receiving certain chemotherapy medications and is hard to treat. Medications commonly used to treat CIPN have limited benefits and may cause significant side effects. A small report showed that topical cannabidiol may help treat neuropathy in patients with diabetes. This study is being done to determine if cannabidiol cream can help improve the symptoms of CIPN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether topical cannabidiol (CBD) improves CIPN, compared to placebo.

II. To evaluate side effects from topical CBD cream use, compared to placebo.

SECONDARY OBJECTIVES:

I. Other measures of neuropathy as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CIPN20 motor subscale, the EORTC QLQ CIPN20 autonomic scale, and the total Common Terminology Criteria for Adverse Events (CTCAE) neuropathy scale.

II. Adverse event profiles will also be assessed using symptom questionnaires and CTCAE version (v)5.0.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients apply cannabidiol cream topically to affected areas twice daily (BID) for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.

ARM II: Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* English speaking
* Cancer diagnosis of any tumor type with chemotherapy-induced neuropathy
* At least 4 out of 10 severity of neuropathy pain and/or tingling
* Stable for at least 7 days prior to registration on medications for neuropathy, if any are being used
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Able to provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* No evidence of residual cancer
* Platelet count > 100,000/mm^3 (following completion of chemotherapy)
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (following completion of chemotherapy)
* Hemoglobin > 11 g/dL (following completion of chemotherapy)
* Serum transaminase (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) =< 1.2 x upper limit of normal (ULN) (following completion of chemotherapy)
* Alkaline phosphatase =< 1.2 x ULN (following completion of chemotherapy)
* Serum creatinine =< 1.2 x ULN (following completion of chemotherapy)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Any medical condition that would prohibit use of a topical cream (skin infection or open wound in the area of the neuropathy)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Pre-existing neuropathy prior to chemotherapy that would confuse the issue of CIPN
* Currently on chemotherapy or received chemotherapy treatment within the prior 3 months
* Use of other cannabis products within 30 days prior to registration
* History of allergy to cannabis products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D. D'Andre, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (9):
- United States (9):
  - Mayo Clinic Health System Albert Lea, Albert Lea, Minnesota
  - Fairview Grand Itasca Clinic and Hospital, Grand Rapids, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Mayo Clinic Health System Mankato, Mankato, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Sanford Thief River Falls, Thief River Falls, Minnesota
  - Sanford Worthington, Worthington, Minnesota

REFERENCES:
- [Derived] D'Andre S, Novotny P, Walters C, Lewis-Peters S, Thome S, Tofthagen CS, Giridhar KV, Loprinzi C. Topical Cannabidiol for Established Chemotherapy-Induced Neuropathy: A Pilot Randomized Placebo-Controlled Trial. Cannabis Cannabinoid Res. 2024 Dec;9(6):e1556-e1564. doi: 10.1089/can.2023.0253. Epub 2024 Jul 17. PMID 39016024
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Cannabidiol, Placebo): Patients apply cannabidiol cream topically to affected areas BID for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.
  >
  > Cannabidiol: Applied topically
  >
  > Placebo Administration: Applied topically
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Arm II (Placebo, Cannabidiol): Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.
  >
  > Cannabidiol: Applied topically
  >
  > Placebo Administration: Applied topically
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
Period: Initial Treatment
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol)
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible | 0 | 1
Period: Crossover
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol)
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Cannabidiol, Placebo): Patients apply cannabidiol cream topically to affected areas BID for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.> > Cannabidiol: Applied topically>
  > Placebo Administration: Applied topically>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Arm II (Placebo, Cannabidiol): Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.> > Cannabidiol: Applied topically>
  > Placebo Administration: Applied topically>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol) | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.3) | 61.3 (10.3) | 62.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Any Prior Cancer Therapy [Count of Participants; unit: Participants] | 20 | 18 | 38
Height (cm) [Mean (Standard Deviation); unit: cm] | 169.1 (8.6) | 170.8 (8.6) | 169.9 (8.5)
Weight (Kg) [Mean (Standard Deviation); unit: Kg] | 87.4 (17.1) | 85.4 (14.8) | 86.5 (15.9)
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 15 | 14 | 29
    1 | 5 | 2 | 7
    2 | 0 | 2 | 2
NCI-CTCAE v5.0 CIPN Grade [Count of Participants; unit: Participants] — Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Death
  Participants
    I | 1 | 1 | 2
    II | 11 | 11 | 22
    III | 3 | 5 | 8
    IV | 5 | 0 | 5
    Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Chemotherapy-induced Peripheral Neuropathy (CIPN) From Baseline
Description: CIPN will be measured by the sensory subscale of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-CIPN20 which is composed of 9 individual items. Each item is scored on a 1-to-4 scale, where 1 means "not at all" and 4 means "very much." Higher scores indicate greater severity of symptoms.
Time Frame: Week 1, week 2, week 3, and week 4
Measure: Mean (95% Confidence Interval); unit: percentage of change in CIPN
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol)
Number analyzed (Participants) | 20 | 17
percentage of change in CIPN
  Week 1 | 147.95 [114.45 to 181.45] | 135.82 [116.34 to 155.30]
  Week 2 | 167.96 [106.64 to 229.28] | 148.45 [120.08 to 176.82]
  Week 3 | 148.83 [113.66 to 184.00] | 140.33 [115.72 to 164.95]
  Week 4 | 181.39 [100.69 to 262.10] | 142.72 [117.75 to 167.69]

2. Secondary Outcome: Change in EORTC QLQ CIPN20 Motor Subscale From Baseline
Description: Motor symptoms of CIPN will be measured by the motor subscale of the EEORTC QLQ-CIPN20 which is composed of 8 individual items. Each item is scored on a 1-to-4 scale, where 1 means "not at all" and 4 means "very much." Higher scores indicate greater severity of symptoms. Will be compared between arms using two-sample, two-sided t-tests. The cannabidiol arm will be compared to the placebo arm. Will construct 95% confidence intervals for the mean difference in sensory neuropathy score between arms. Repeated measures mixed models will be applied to the sensory scores over all time points to determine longitudinal effects and to adjust for confounding factors. Graphical results will include profile plots over time, stream plots of individual changes over time, and forest plots of the 95% confidence intervals by arm.
Time Frame: Week 1, week 2, week 3, and week 4
Measure: Mean (95% Confidence Interval); unit: percentage of change in EORTC
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol)
Number analyzed (Participants) | 20 | 17
percentage of change in EORTC
  Week 1 | 129.79 [107.30 to 152.27] | 114.11 [99.34 to 128.89]
  Week 2 | 135.63 [108.05 to 163.21] | 131.13 [105.68 to 156.57]
  Week 3 | 126.09 [104.67 to 147.50] | 121.61 [103.249 to 139.974]
  Week 4 | 134.85 [107.531 to 162.158] | 123.26 [104.14 to 142.37]

3. Secondary Outcome: Change in EORTC QLQ CIPN20 Autonomic Scale From Baseline
Description: Autonomic nervous system symptoms related to CIPN will be measured by the autonomic subscale of the EEORTC QLQ-CIPN20 which is composed of 3 individual items answered on a 4-point scale ranging from "not at all' to "very much." . Higher scores indicate more severe symptoms. Will be compared between arms using two-sample, two-sided t-tests. The cannabidiol arm will be compared to the placebo arm. Will construct 95% confidence intervals for the mean difference in sensory neuropathy score between arms. Repeated measures mixed models will be applied to the sensory scores over all time points to determine longitudinal effects and to adjust for confounding factors. Graphical results will include profile plots over time, stream plots of individual changes over time, and forest plots of the 95% confidence intervals by arm.
Time Frame: Week 1, week 2, week 3, and week 4
Measure: Mean (95% Confidence Interval); unit: percentage of change in EORTC
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol)
Number analyzed (Participants) | 20 | 17
percentage of change in EORTC
  Week 1 | 110.88 [91.99 to 129.76] | 99.59 [91.59 to 107.58]
  Week 2 | 123.91 [106.78 to 141.04] | 100.85 [93.20 to 108.50]
  Week 3 | 112.07 [97.92 to 126.52] | 100.55 [89.93 to 111.17]
  Week 4 | 120.71 [103.52 to 137.91] | 104.34 [95.30 to 113.37]

4. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Incidence of AEs will be reported per arm, assessed using Common Terminology Criteria (CTCAE) version 5.0.
Time Frame: Up to 14 days for each part of a sequence
Measure: Count of Participants; unit: Participants
Groups:
- Arm I Crossover (Cannabidiol, Placebo): Patients apply cannabidiol cream topically to affected areas BID for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.
  Cannabidiol: Applied topically
  Placebo Administration: Applied topically
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Arm II Crossover (Placebo, Cannabidiol): Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.
  Cannabidiol: Applied topically
  Placebo Administration: Applied topically
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol) | Arm I Crossover (Cannabidiol, Placebo) | Arm II Crossover (Placebo, Cannabidiol)
Number analyzed (Participants) | 20 | 20 | 19 | 17
Participants
  Spinal fracture | 1 | 0 | 0 | 0
  Back pain | 1 | 0 | 0 | 0
  Hypotension | 1 | 0 | 0 | 0

5. Secondary Outcome: Incidence of Grade 3 or Higher Adverse Events
Description: Will be assessed using symptom questionnaires and CTCAE version 5.0. Will compare the maximum (worst) values between arms. Fisher's exact tests will be used to compare incidence rates and Wilcoxon rank-sum tests will be used to compare maximum values between arms.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Arm I Crossover (Cannabidiol, Placebo): Patients apply cannabidiol cream topically to affected areas BID for 14 days. Patients then apply placebo cream topically to affected areas BID for 14 days.
  >
  > Cannabidiol: Applied topically
  >
  > Placebo Administration: Applied topically
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Arm II Crossover (Placebo, Cannabidiol): Patients apply placebo cream topically to affected areas BID for 14 days. Patients then apply cannabidiol cream topically to affected areas BID for 14 days.
  >
  > Cannabidiol: Applied topically
  >
  > Placebo Administration: Applied topically
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol) | Arm I Crossover (Cannabidiol, Placebo) | Arm II Crossover (Placebo, Cannabidiol)
Number analyzed (Participants) | 20 | 20 | 19 | 17
Participants
  Grade 3 | 2 | 0 | 0 | 0
  Grade 4+ | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days
Groups:
- Arm I Crossover (Cannabidiol, Placebo); Arm II Crossover (Placebo, Cannabidiol): Questionnaire Administration: Ancillary studies
Arm/Group | Arm I (Cannabidiol, Placebo) | Arm II (Placebo, Cannabidiol) | Arm I Crossover (Cannabidiol, Placebo) | Arm II Crossover (Placebo, Cannabidiol)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20 | 0/19 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cannabidiol, Placebo) (N=20) | Arm II (Placebo, Cannabidiol) (N=20) | Arm I Crossover (Cannabidiol, Placebo) (N=19) | Arm II Crossover (Placebo, Cannabidiol) (N=17)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT05388058/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT05388058/ICF_001.pdf